CLINICAL TRIAL: NCT05440851
Title: Platform of Randomized Adaptive Clinical Trials in Critical Illness
Acronym: PRACTICAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-5940
Record Dates: First submitted 2021-11-10; First posted 2022-07-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Insufficiency; Extracorporeal Membrane Oxygenation Complication; Mechanical Ventilation Pressure High
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Fludrocortisone; Airway Extubation; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: While blinding of treatment allocation is an important mechanism for mitigating bias, the nature of acute hypoxemic respiratory failure and the complexity of interventions to be tested in PRACTICAL may make it difficult to blind treatment allocation in some cases. Blinded allocation will be implemented where possible.
  Where possible, clinical outcomes will be collected by research personnel who are masked to randomized treatment assignment. Even where research personnel cannot be blinded to treatment assignment, bias arising will be mitigated by selection of relatively objective endpoints not easily influenced by knowledge of treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Ultra-protective ventilation facilitated by extracorporeal carbon dioxide removal. (Other): Patients randomized to the this intervention group will receive VV-ECMO with the ventilator set to minimize driving pressure and respiratory rate for ultra-protective ventilation.
  Interventions: Other: Ultra-Protective Ventilation Facilitated by Extracorporeal Support; Other: Lung-Protective Ventilation (LPV); Other: VV ECMO-facilitated strategy of earlier awakening, extubation and rehabilitation
- Invasive Mechanical Ventilation (IMV) Strategies domain (Other): Patients on invasive mechanical ventilation in the low elastance, high elastance, and ECLS states will be randomized to minimum of one of two mechanical ventilation interventions (including conventional lung-protective ventilation as a control group). Most sites will randomize patients to two arms (one of which is the control group, LPV). A subset of sites will randomize patients to all three or four arms.
  Interventions: Other: Lung-Protective Ventilation (LPV); Other: Driving Pressure-Limited Ventilation (DPL); Other: Lung- and Diaphragm-Protective Ventilation and Sedation (LDPVS); Other: Electrical impedance tomography (EIT)
- The Corticosteroid Early and Extended (CORT-E2) Randomized Controlled Trial domain (Other): Patients with acute hypoxemic respiratory failure (AHRF) requiring invasive or non-invasive respiratory support will be randomized in the Early Cohort to receive corticosteroid or usual care without corticosteroids. Patients treated with corticosteroids who still require invasive or non-invasive respiratory support after 10 days will be randomized in the Extended Cohort to extending corticosteroid use or stopping corticosteroids after 10 days.
  Interventions: Drug: Early Cohort corticosteroid dose; Drug: Extended Cohort corticosteroid dose; Drug: Usual care without routine corticosteroids; Drug: Usual care without extending corticosteroids
- The Nebulized Furosemide for the Treatment of Pulmonary Inflammation (FAST-3) domain (Other): Patients with Respiratory Failure Secondary to Pulmonary Infection.
  Interventions: Drug: 4 mL of nebulized 0.9% saline minutes every 6 hours over 30 minutes every 6 hours.; Drug: 40 mg of nebulized furosemide in 4 mL of saline nebulized over 30 minutes every 6 hours
- The Invasive Mechanical Ventilation Strategies in Venovenous-Extracorporeal Life Support (IMV-ECLS) (Other): Patients with acute hypoxemic respiratory failure receiving extracorporeal life support will be randomized to one of three positive end-expiratory pressure (PEEP) strategies.
  Interventions: Other: PEEP-20; Other: PEEP-AOP; Other: PEEP-10
- The Fludrocortisone in Acute Hypoxemic Respiratory Failure with Airspace Disease (FLUDRO-1) domain (Other): Patients with acute hypoxemic respiratory failure with airspace disease will be randomized to usual care with or without fludrocortisone.
  Interventions: Drug: Usual care with fludrocortisone; Drug: Usual care without fludrocortisone
- VV ECMO-facilitated strategy of earlier awakening, extubation and rehabilitation (Other): Patients with acute hypoxemic respiratory failure in the high elastance state will be randomized to ultra-protective ventilation facilitated by extracorporeal carbon dioxide removal or to VV ECMO-facilitated strategy of earlier awakening, extubation and rehabilitation or to conventional lung-protective ventilation.
  Interventions: Other: Ultra-Protective Ventilation Facilitated by Extracorporeal Support; Other: Lung-Protective Ventilation (LPV); Other: VV ECMO-facilitated strategy of earlier awakening, extubation and rehabilitation
- Evaluating Subphenotypes in Immunocompromized Patients with ARF (ESCAPE) Domain (Other): We will conduct a prospective, multicenter, observational study (no treatment arm is involved) in 7 ICUs in Canada over 3 years. We will include adult patients (≥18 years) admitted to the ICU with AHRF who have an underlying immunocompromised condition.
  Biomarker Collection: Samples for serum biomarkers will be collected within 24 hours of fulfilling inclusion criteria, on days 0, 3 and 7. We will collect biomarkers associated with inflammatory conditions, epithelial injury, endothelial dysfunction and coagulation abnormalities - which have been shown to characterize lung injury or critical illness.
  Data Collection: We will collect demographic, comorbidity, immunocompromised defining condition, clinical, respiratory physiology, and serum biomarker data for each patient.
  Interventions: Other: no treatment / intervention arm is involved
- Inspiratory Muscle Training in Patients Receiving Ongoing Mechanical Ventilation (IMPROV) Domain (Other): This domain studies inspiratory muscle training (IMT) during and after mechanical ventilation in patients with acute hypoxemic respiratory failure (AHRF).
  Interventions: Other: Usual care; Other: Early Routine IMT

INTERVENTIONS:
Other: Ultra-Protective Ventilation Facilitated by Extracorporeal Support — Patients randomized to this intervention group will receive VV-ECMO with the ventilator set to minimize driving pressure and respiratory rate for ultra-protective ventilation.
  Arms: Ultra-protective ventilation facilitated by extracorporeal carbon dioxide removal.; VV ECMO-facilitated strategy of earlier awakening, extubation and rehabilitation
Other: Lung-Protective Ventilation (LPV) — Patients randomized to LPV will receive standard of care lung-protective ventilation with conventional limits on tidal volume and plateau airway pressure.
  Arms: Invasive Mechanical Ventilation (IMV) Strategies domain; Ultra-protective ventilation facilitated by extracorporeal carbon dioxide removal.; VV ECMO-facilitated strategy of earlier awakening, extubation and rehabilitation
Other: Driving Pressure-Limited Ventilation (DPL) — Patients randomized to DPL will receive mechanical ventilation set to maintain a safe limit on driving pressure and plateau airway pressure, without less for the tidal volume.
  Arms: Invasive Mechanical Ventilation (IMV) Strategies domain
Other: Lung- and Diaphragm-Protective Ventilation and Sedation (LDPVS) — Patients randomized to LDPVS will have ventilation and sedation adjusted to maintain lung-distending pressure and respiratory effort in a safe target range.
  Arms: Invasive Mechanical Ventilation (IMV) Strategies domain
Drug: Early Cohort corticosteroid dose — Patients randomized to receive corticosteroids will receive dexamethasone 20mg daily for 5 days and then 10mg for an additional 5 days, for a total of 10 days from the time of randomization (or until ICU discharge or death, whichever comes first); after 10 days dexamethasone will be stopped without a taper.
  Arms: The Corticosteroid Early and Extended (CORT-E2) Randomized Controlled Trial domain
Drug: Extended Cohort corticosteroid dose — Patients randomized to receive extended corticosteroids will receive dexamethasone 10mg for an additional 10 days. At the end of the additional 10 days (day 20 of corticosteroids), the dexamethasone dose will be halved to 5mg for another 5 days (to reduce the risk of adrenal insufficiency) and then stopped (a total of 25 days or until ICU discharge or death, whichever comes first).
  Arms: The Corticosteroid Early and Extended (CORT-E2) Randomized Controlled Trial domain
Drug: Usual care without routine corticosteroids — Patients randomized to this arm will be managed according to usual care. They will receive corticosteroids only if prescribed by the clinician.
  Arms: The Corticosteroid Early and Extended (CORT-E2) Randomized Controlled Trial domain
Drug: Usual care without extending corticosteroids — Corticosteroids will stop after 10 days. Other management will be according to usual care. Patients will receive corticosteroids only if prescribed by the clinician.
  Arms: The Corticosteroid Early and Extended (CORT-E2) Randomized Controlled Trial domain
Drug: Usual care with fludrocortisone — Best practice standard of care prescribed by treating team + fludrocortisone 50μg enterally daily for 7 days.
  Arms: The Fludrocortisone in Acute Hypoxemic Respiratory Failure with Airspace Disease (FLUDRO-1) domain
Drug: Usual care without fludrocortisone — Best practice standard of care prescribed by treating team without fludrocortisone. After randomization, if a clinical indication develops for fludrocortisone as part of standard of care, administration of fludrocortisone is not prohibited. Any fludrocortisone administered to participants in the control arm will be documented.
  Arms: The Fludrocortisone in Acute Hypoxemic Respiratory Failure with Airspace Disease (FLUDRO-1) domain
Drug: 4 mL of nebulized 0.9% saline minutes every 6 hours over 30 minutes every 6 hours. — 4 mL of nebulized 0.9% saline minutes every 6 hours over 30 minutes every 6 hours.
  Arms: The Nebulized Furosemide for the Treatment of Pulmonary Inflammation (FAST-3) domain
Drug: 40 mg of nebulized furosemide in 4 mL of saline nebulized over 30 minutes every 6 hours — 40 mg of nebulized furosemide in 4 mL of saline nebulized over 30 minutes every 6 hours
  Arms: The Nebulized Furosemide for the Treatment of Pulmonary Inflammation (FAST-3) domain
Other: PEEP-20 — fixed high positive end-expiratory pressure at 20 cmH2O
  Arms: The Invasive Mechanical Ventilation Strategies in Venovenous-Extracorporeal Life Support (IMV-ECLS)
Other: PEEP-AOP — positive end-expiratory pressure set according to airway opening pressure
  Arms: The Invasive Mechanical Ventilation Strategies in Venovenous-Extracorporeal Life Support (IMV-ECLS)
Other: PEEP-10 — fixed lower positive end-expiratory pressure at 10 cmH2O
  Arms: The Invasive Mechanical Ventilation Strategies in Venovenous-Extracorporeal Life Support (IMV-ECLS)
Other: VV ECMO-facilitated strategy of earlier awakening, extubation and rehabilitation — Patients randomized to this intervention group will receive VV-ECMO where the sedation will be reduced and the ventilator will will be adjusted to facilitate spontaneous breathing.
  Arms: Ultra-protective ventilation facilitated by extracorporeal carbon dioxide removal.; VV ECMO-facilitated strategy of earlier awakening, extubation and rehabilitation
Other: Electrical impedance tomography (EIT) — Patients randomized to EIT will have PEEP titration compared via the Overdistension Collapse Intercept (ODCL) versus that obtained using a standard high PEEP table.
  Arms: Invasive Mechanical Ventilation (IMV) Strategies domain
Other: no treatment / intervention arm is involved — This trial is a prospective, multicenter, observational study (no treatment arm is involved).
  Arms: Evaluating Subphenotypes in Immunocompromized Patients with ARF (ESCAPE) Domain
Other: Usual care — Patients will be treated according to usual care.
  Arms: Inspiratory Muscle Training in Patients Receiving Ongoing Mechanical Ventilation (IMPROV) Domain
Other: Early Routine IMT — * Training commences once patients meet readiness to wean criteria
  * 3 sets of 10 breaths, delivered twice daily using a device placed at the airway opening to apply an external resistive pressure load, until hospital discharge, death, or day 45 after randomization, whichever occurs first.
  * Device load will initially be set to 30% of the MIP.
  * Device load will be titrated upward (in increments of 5-10% of MIP, to a maximum of 60% of MIP) as needed to achieve a modified Borg dyspnea score of 7/10 or visible accessory muscle use.
  Arms: Inspiratory Muscle Training in Patients Receiving Ongoing Mechanical Ventilation (IMPROV) Domain

SUMMARY:
PRACTICAL is a randomized multifactorial adaptive platform trial for acute hypoxemic respiratory failure (AHRF). This platform trial will evaluate novel interventions for patients with AHRF across a range of severity states (i.e., not intubated, intubated with lower or higher respiratory system elastance, requiring extracorporeal life support) and across a range of investigational phases (i.e., preliminary mechanistic trials, full-scale clinical trials). AHRF is a common and life-threatening clinical syndrome affecting millions globally every year. Patients with AHRF are at high risk of death and long-term morbidity. Patients who require invasive mechanical ventilation are at risk of ventilator-induced lung injury and ventilator-induced diaphragm dysfunction. New treatments and treatment strategies are needed to improve outcomes for these very ill patients.

Utilizing advances in Bayesian adaptive trial design, the platform will facilitate efficient yet rigorous testing of new treatments for AHRF, with a particular focus on mechanical ventilation strategies and extracorporeal life support techniques as well as pharmacological agents and new medical devices.

The platform is designed to enable evaluation of novel interventions at a variety of stages of investigation, including pilot and feasibility trials, trials focused on mechanistic surrogate endpoints for preliminary clinical evaluation, and full-scale clinical trials assessing the impact of interventions on patient-centered outcomes.

Interventions will be evaluated within therapeutic domains. A domain is defined as a set of interventions that are intended to act on specific mechanisms of injury using different variations of a common therapeutic strategy. Domains are intended to function independently of each other, allowing independent evaluation of multiple therapies within the same patient.

Once feasibility is established, Bayesian adaptive statistical modelling will be used to evaluate treatment efficacy at regular interim adaptive analyses of the pre-specified outcomes for each intervention in each domain. These adaptive analyses will compute the posterior probabilities of superiority, futility, inferiority, or equivalence for pre-specified comparisons within domains. Each of these potential conclusions will be pre-defined prior to commencing the intervention trial. Decisions about trial results (e.g., concluding superiority or equivalence) will be based on pre-specified threshold values for posterior probability. The primary outcome of interest, the definitions for superiority, futility, etc. (i.e., the magnitude of treatment effect) and the threshold values of posterior probability required to reach conclusions for superiority, futility etc., will vary from intervention to intervention depending on the phase of investigation and the nature of the intervention being evaluated. All of these parameters will be pre-specified as part of the statistical design for each intervention trial.

In general, domains will be designed to evaluate treatment effect within four discrete clinical states: non-intubated patients, intubated patients with low respiratory system elastance (<2.5 cm H2O/(mL/kg)), intubated patients with high respiratory system elastance (≥2.5 cm H2O/(mL/kg)), and patients requiring extracorporeal life support. Where appropriate, the model will specify dynamic borrowing between states to maximize statistical information available for trial conclusions. In this perpetual trial design, different interventions may be added or dropped over time.

Where possible, the platform will be embedded within existing data collection repositories to enable greater efficiency in outcome ascertainment. Standardized systems for acquiring both physiological and biological measurements are embedded in the platform, to be acquired at sites with appropriate training, expertise, and facilities to collect those measurements.

DETAILED DESCRIPTION:
EXPAND-ECLS domain: The EXPAND-ECLS pilot trial is a multi-center, randomized, open-label, feasibility trial, embedded as a domain within the PRACTICAL platform trial. The ULTIMATE arm of this domain will evaluate the effect of ultra-low intensity ventilation facilitated by CO2 removal through VV-ECMO versus best current conventional ventilation on all-cause hospital mortality among patients with early moderate-severe AHRF with high respiratory system elastance receiving potentially injurious mechanical ventilation. The PROACTIVE arm of this domain will evaluate the effect of ECMO-facilitated strategy of earlier awakening, extubation, and rehabilitation versus best current conventional ventilation on all-cause hospital mortality among patients with early moderate-severe AHRF with high respiratory system elastance receiving potentially injurious mechanical ventilation.

Invasive Mechanical Ventilation (IMV) Strategies domain: The IMV Strategies domain will evaluate multiple novel invasive ventilation strategies in comparison to conventional lung-protective ventilation in patients with acute hypoxemic respiratory failure (AHRF). Multiple approaches to mechanical ventilation are used, and the optimal approach is unknown. An efficient strategy to identify the best strategy is to compare multiple potential approaches simultaneously to determine more rapidly (a) which interventions are least effective (and should be dropped), and (b) which interventions result in the best outcomes for patients. In the current domain design, we will compare the current recommended ventilation strategy to two new approaches: a strategy that targets lung-inflating (driving) pressure instead of lung-inflating (tidal) volume, and a strategy that aims to maintain an optimal level of breathing effort to prevent diaphragm atrophy and injury while maintaining safe lung-inflating pressures.

CORT-E2 domain: The Corticosteroid Early and Extended (CORT-E2) Trial is a phase III, multicentre Bayesian randomized controlled trial (RCT), which includes two cohorts within the domain; one examining the role of early corticosteroids as compared to not extending in persisting AHRF due to COVID or non-COVID (Extended Cohort).

ESCAPE domain: Evaluating Subphenotypes in Immunocompromized Patients with ARF (ESCAPE) Domain is a prospective, multicentre observational cohort study, to identify subphenotypes across immunocompromised patients with acute hypoxemic respiratory failure (AHRF) using clinical characteristics and biomarkers. This study will prospectively collect biomarkers at the onset of AHRF which will allow us to characterize the underlying pathophysiology of AHRF with better precision.

FLUDRO domain: The Fludrocortisone in Acute Hypoxemic Respiratory Failure with Airspace Disease (FLUDRO-1) domain is a phase II I trial. The trial aims to provide direct clinical evidence to resolve a critical long-standing question regarding the use of steroids in the treatment of AHRF with airspace disease.

FAST-3 domain: The Nebulized Furosemide for the Treatment of Pulmonary Inflammation in Patients with Respiratory Failure Secondary to Pulmonary Infection domain is a phase III trial. It aims to use nebulized furosemide as supportive therapy to improve Advanced Respiratory Support (ARS) free days up to day 28 in critically ill patients with AHRF.

IMV-ECLS domain: The Invasive Mechanical Ventilation Strategies in Venovenous-Extracorporeal Life Support (PRESSURE; Positive Pressure to Maintain Lung Recruitment during Extracorporeal Life Support for Acute Hypoxemic Respiratory failure) is a pilot and feasibility trial. It aims to identify which positive end-expiratory pressure (PEEP) strategies improve lung function in patients with AHRF supported by ECLS.

IMPROV domain: The Inspiratory Muscle Training in Patients Receiving Ongoing Mechanical Ventilation is a pilot and feasibility RCT. It is designed to establish the feasibility of a definitive RCT of inspiratory muscle training to accelerate recovery from AHRF.

ELIGIBILITY:
PRACTICAL Platform Inclusion Criteria:

1. Acute hypoxemic respiratory failure meeting all of the following criteria;

   1. New or worsening respiratory symptoms developing within 2 weeks prior to the onset of need for oxygen or respiratory support
   2. Receiving any of the following types of oxygen or respiratory support for at least 4 hours prior to the time of randomization; supplemental oxygen at 10 L/min or higher, high flow nasal oxygen (at any flow rate), invasive ventilator support, extra-corporeal life support (ECLS), or non-invasive ventilator support
   3. Minimum FiO2 ≥ 0.40 (for venturi mask, high flow nasal cannula, or invasive or non-invasive ventilation) or oxygen flow rate ≥10 L/min on face mask for at least 4 hours at the time of evaluation for eligibility unless already on extra-corporeal life support
2. Age ≥ 18 years
3. Hypoxemia not primarily attributable to acute heart failure, fluid overload, or pulmonary embolism (PE)

PRACTICAL Platform Exclusion Criteria:

1. Extubation is planned or anticipated on the day of screening
2. ICU discharged is planned or anticipated on the day of screening
3. If the patient is moribund and deemed unlikely to survive 24 hours (as determined by the clinical team)
4. If the patient is being transitioned to a fully palliative philosophy of care

EXPAND-ECLS Domain Inclusion Criteria:

1. Receiving invasive Endotracheal mechanical ventilation for ≤ 72 hours.5 days
2. Early Moderate-severe hypoxemic respiratory failure with a PaO2/FiO2≤150200 mmHg for at least 6 hours

EXPAND-ECLS Domain Exclusion Criteria:

1. Patients over 70 years of age.
2. Currently receiving any form of ECLS (e.g., Venovenous, venoarterial, or hybrid configuration).
3. Chronic hypercapnic respiratory failure defined as PaCO2 > 60 mmHg in the outpatient setting.
4. Home mechanical ventilation (non-invasive ventilation or via tracheotomy) except for CPAP/BiPAP used solely for sleep-disordered breathing.
5. Actual body weight exceeding 1 kg per centimeter of height.
6. More than 48 hours have passed since meeting inclusion criteria.
7. Severe hypoxemia with PaO2/FiO2 < 80mmHg for > 6 hours at time of screening.
8. Severe hypercapnic respiratory failure with pH < 7.25 and PaCO2 > 60 mmHg for > 6 hours at time of screening.
9. Expected mechanical ventilation duration < 48 hours at time of screening.
10. Confirmed diffuse alveolar hemorrhage from vasculitis.
11. Contraindications to limited anticoagulation (e.g., active GI bleeding, bleeding diathesis).
12. Previous hypersensitivity/anaphylactic reaction to heparin or heparin-induced thrombocytopenia
13. Neurologic conditions at risk for or undergoing treatment for intracranial hypertension
14. Underlying illness with life expectancy < 1 year
15. Pregnancy (due to unknown effects of PaCO2 changes on placental blood flow)
16. Respiratory failure known or suspected to be caused by COVID-19.

IMV Domain Inclusion Criteria:

1. Intubated patients, not on ECLS, with low normalized respiratory elastance (<2.5 cm H2O/(ml/kg predicted body weight)) at the time of eligibility assessment OR
2. Intubated patients, not on ECLS, with high normalized respiratory system elastance (≥2.5 cm H2O/(ml/kg predicted body weight)) at the time of eligibility assessment OR
3. FOR STUDY SITES PARTICIPATING IN THE LDPVS INTERVENTION: Patient is on ECLS at the time of eligibility assessment. Note: Patients in this state are only eligible for the LPV or LDPVS intervention
4. FOR STUDY SITES PARTICPATING IN THE EIT INTERVENTION: PaO2/FiO2 (if available) < 200 mm Hg at randomization. If PaO2/FiO2 has not been measured, SpO2 = 97% on FiO2 =60%.

IMV Domain Exclusion Criteria:

1. PaO2/FiO2 >300 mm Hg or (S/F >250, if PaO2/FiO2 has not been measured) at the time of randomization 2. Chronic hypercapnic respiratory failure defined as PaCO2>60mmHg in the outpatient setting 3. Home mechanical ventilation (non-invasive ventilation or via tracheotomy), not including nocturnal CPAP applied by nasal or face mask or home tracheotomy if not ventilated 4. Severe hypoxemia with PaO2/FiO2<80mmHg for >6 consecutive hours at the time of randomization 5. Severe hypercapnic respiratory failure with pH<7.25 and PaCO2>60mmHg for >6 consecutive hours at the time of randomization 6. Anticipated duration of mechanical ventilation is <48 hours from the time of screening 7. Duration of mechanical ventilation during current ICU admission is >72 hours 8. Previously diagnosed neuromuscular disorder 9. Current diagnosis of severe acute brain injury (e.g. ischemic or hemorrhagic stroke, traumatic brain injury) with Glasgow Coma Scale ≤ 8 10. Baseline weight prior to or at hospital admission less than 35 kilograms 11. Receiving extracorporeal life support without continuous invasive mechanical ventilatory support

CORT-E2 Domain Early Cohort Inclusion Criteria

1. Within 72 hours of admission to an ICU
2. New unilateral or bilateral airspace disease

CORT-E2 Domain Early Domain Exclusion Criteria

1. Receiving only low flow oxygen therapy less than or equal to 15L/min
2. Corticosteroid use during the 14 days prior to screening
3. Existing indication for corticosteroids
4. High suspicion for/or confirmed COVID infection
5. Acute traumatic brain injury during the index hospital admission
6. Allergy to dexamethasone

CORT-E2 Domain Extended Cohort Inclusion Criteria

1. Are admitted to an ICU
2. Have already received 10 days of corticosteroid specifically for acute respiratory failure, this will include patients: (a) randomized to corticosteroid arm in Early Cohort, (b) patients with COVID receiving corticosteroids as standard of care , (c) and others who have received corticosteroids for AHRF
3. Ongoing AHRF requiring HFNC, NIV (continuous positive airway pressure [CPAP] or bilevel) or invasive ventilation

CORT-E2 Domain Extended Cohort Exclusion Criteria

1. An alternate indication for ongoing corticosteroids
2. Acute traumatic brain injury this hospital admission

FLUDRO Domain Inclusion Criteria

1. Within 72 hours of admission to an ICU

FLUDRO Domain Exclusion Criteria

1. Known hypersensitivity to fludrocortisone
2. An inability to receive fludrocortisone due to lack of enteral access
3. An indication to prescribe fludrocortisone for a reason that is unrelated to a current episode of pneumonia or acute respiratory failure, such as Addison's disease
4. Belief of the treating clinical team that study participation would not be in the best interest of the patient

FAST-3 Domain Inclusion Criteria (must meet all 3 of the following)

1. Patient is in a PRACTICAL eligible platform state and requires advanced respiratory support (ARS) defined as one of the following:

   a. Invasive mechanical ventilation with FiO2 > 40% b. Non-Invasive Ventilation (> 4 hours consecutively with FiO2 > 40%) defined as: i. CPAP or BiPAP (any settings or interface) ii. HFNC (flow > 40 liter per minute)
2. PaO2/FiO2 < 300 mm Hg or SpO2/FiO2 < 315 (if PaO2/FiO2 unavailable due to lack of arterial blood gas at the time of screening). For SpO2/FiO2, criteria are SpO2 ≤ 97% on FiO2 ≥ 40% on both of the 2 hours immediately preceding eligibility assessment. If an arterial blood gas can be obtained, then a PaO2/FiO2 ratio is preferable.
3. Patient commenced advanced respiratory support < 48 hours prior to randomization.

FAST-3 Domain Exclusion Criteria

1. Patient commenced advanced respiratory support > 48 hours to time of randomization.
2. Known history of severe chronic pulmonary disease e.g., pre-infection requirement for home oxygen therapy or presence of chronic hypercapnia (PaCO2 > 60 mmHg); mild - moderate disease is still eligible in the absence of chronic hypercapnia or need for chronic oxygen therapy.
3. Currently enrolled in another trial studying investigational anti-inflammatory therapy, excluding established treatments used in clinical practice such as corticosteroids.
4. Known allergy to furosemide or sulfonamide drugs. If the patient is allergic to sulfonamide drugs but has received in the past or is currently receiving furosemide without incident, they can be enrolled since cross-reactivity between furosemide and sulfonamide agents is rare.

ESCAPE Domain Inclusion Criteria

1. Patients with severe AHRF who have an underlying immunocompromised condition
2. Within 48 hours of fulfilling the AHRF inclusion criteria as well as PaO2/FiO2 <300 or a SaO2/FiO2 < 315 on non-invasive respiratory support (venturi mask, non-invasive ventilation or high flow nasal oxygen as per the FiO2 requirements above) or invasive ventilation.

Patients may be enrolled from the wards or ICU.

Immunocompromised patients include:

1. Any patients requiring long term (>30 days) corticosteroids (>20 mg/day),
2. Any patients receiving non-corticosteroid immunosuppressive medications within the prior 3 months,
3. Acquired or inherited immunodeficiency syndrome,
4. Recipients of solid organ transplant,
5. Active hematologic malignancy (diagnosis or receiving treatment within prior 6 months),
6. Active solid tumor (diagnosis or receiving treatment within the prior 6 months) or
7. Any patients who have undergone allogeneic or autologous hematopoietic cell transplant in the prior 6 months (HCT).

   ESCAPE Domain Exclusion Criteria 1. Patients whom are deemed palliative.

   IMV-ECLS Domain Inclusion Criteria

   1. Patients with AHRF (as defined in platform inclusion criteria #1 above) who have been consented for cannulation for VV-ECLS or who have been initiated on VV-ECLS within 6 hours at the time of randomization

   IMV-ECLS Domain Exclusion Criteria 1. Patients receiving ECLS for the primary intention of extracorporeal CO2 removal 2. Patients expected to be liberated from ECLS within <24 hours 3. History of recent pneumothorax or pneumomediastinum (<3 months at the time of eligibility assessment/randomization) 4. Patients receiving ECLS for the primary intention of bridge to lung transplantation (at the time of eligibility assessment/randomization)

   IMPROV Domain Inclusion Criteria

   1. Patients receiving invasive mechanical ventilation for AHRF as defined by the PRACTICAL platform trial criteria above.

   2. Within 7 calendar days of intubation

   IMPROV Domain Exclusion Criteria
   1. Patient is expected to be liberated from mechanical ventilation within 24 hours
   2. Known or suspected chronic hypercapnic respiratory failure defined as PaCO2>60mmHg in the outpatient setting
   3. Home mechanical ventilation (non-invasive ventilation or via tracheotomy), not including nocturnal CPAP applied by nasal or face mask or home tracheotomy if not ventilated
   4. Known pneumothorax or pneumomediastinum without chest tube placement sustained during current ICU admission* (re-confirm immediately prior to randomization)
   5. Patient is admitted primarily for acute brain injury (stroke, traumatic brain injury, etc.)
   6. Previously diagnosed chronic neuromuscular disorder
   7. Patient has an implantable cardiac defibrillator or pacemaker
   8. Planned to be transferred to another hospital before ICU discharge
   9. Already receiving a regimen of inspiratory muscle training using external resistive device or diaphragm neurostimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6250 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
EXPAND-ECLS domain - determine the feasibility of recruiting 100 patients over 2 years of active enrolment, as well as assess the rate of participant recruitment and understand the barriers to enrollment. | 2 years of active site enrollment.
  Record total number of patients randomized, total number of patients eligible yet not randomized, and the number of active randomizing sites on a monthly basis. This will include evaluating the validity and appropriateness of inclusion and exclusion criteria, trial acceptability, and reasons for lack of consent or withdrawal.
FLUDRO-1 and IMV domains - ventilator-free days to day 28 in DPL vs LPV (DRIVE RCT) | Day 28 post randomization
  Ventilator-free days to day 28 is computed as an ordinal scale ranging between -1 to 28. Patients who die in hospital will be assigned a value of -1. Otherwise the endpoint will be computed from the number of days alive and free of ventilation in the period between the day the patient is liberated from mechanical ventilation and day 28.
IMV domain - adherence to LDPVS management (LANDMARK RCT) | Day 28
  Adherence to LDPVS management will be measured in terms of the proportion of protocol-specified measurements of respiratory effort that are on target during the intervention period.
IMV domain - probability of achieving and maintaining lung- and diaphragm-protective targets during mechanical ventilation (LANDMARK RCT) | Day 28
  Lung- and diaphragm-protective targets are defined as an estimated dynamic trans pulmonary driving pressure ≤23 cm H2O and a Pocc value between -6 to -20 cm H2O.
IMV domain - protocol adherence (EIT intervention) | Day 9
  Protocol adherence will be measured as a binary outcome daily, while patients are receiving EIT. The target protocol adherence across patients is ≥80%.
CORT-E2 domain - 60-day mortality from the day of randomization | Day 60
FLUDRO-1 domain - Successful enrollment of participants | 18-month enrolment period across three platform trials (PRACTICAL, REMAP-CAP and ATTACC-CAP)
  Protocol adherence: e.g., proportion of participants randomized to fludrocortisone who received the study drug as specified in the protocol; Consent rate; Early withdrawal from domain intervention; Outcome completeness
FAST-3 domain - Advanced respiratory support free days | Day 28
  Advanced respiratory support free days (ARSFDs) to day 28, a composite outcome including mortality and requirement for respiratory support
IMV-ECLS domain - feasibility of enrollment and protocol adherence | For feasibility of enrollment: 2 years of active site enrollment; For protocol adherence, these will be evaluated at 7 days (once the intervention period ends)
  Feasibility of enrollment defined as ≥1 patient enrolled per month per site. Protocol adherence defined as ≥90% of patients initiated on assigned PEEP strategy within 6 hours of ECLS cannulation and ≥90% average protocol adherence across participants.
ESCAPE domain - 28-day all-cause mortality | 28-day
IMPROV domain - recruitment rate, protocol adherence, and vital status | Throughout trial enrollment for recruitment rate and protocol adherence, and up to day 90 for vital status.
  ≥0.75 patients randomized per site per month, Protocol adherence defined as > 80% across participants, and ≥89% ascertainment of vital status and days alive and at home at day 90.

SECONDARY OUTCOMES:
To assess adherence to our explicit mechanical ventilation protocols. | 48 hours
  Adherence to protocol defined as >80% of patients having <20% of monitored values determined to be major protocol deviations.
To measure and understand the reasons for crossovers in each group | 2 years
  Success for lack of crossovers defined as <10% of crossovers between groups (when not allowed by protocol) in either direction.
Duration of mechanical ventilation during index ICU admission | Until ICU discharge, typically within 28 days
  Measured in CORT-E2, IMV, IMV-ECLS and EXPAND-ECLS domains
Mortality at other endpoints | ICU discharge, hospital discharge, day 30, 180 days for CORT-E2, IMV, IMV-ECLS, and EXPAND-ECLS domains. For ESCAPE, Hospital mortality at 60 days and at 6-months. For FAST-3, all-cause mortality at 60 days post enrollment. For IMPROV at day 90.
  Measured in CORT-E2, ESCAPE, FAST-3, IMV, IMV-ECLS, IMPROV and EXPAND-ECLS domains
Vital status | Day 90 and at 6 months
  Measured in IMPROV domain
Duration of ICU admission | Until ICU discharge, typically within 28 days
  Measured in FAST-3, IMV, IMV-ECLS and EXPAND-ECLS domains
Hospital length of stay | Until hospital discharge, assessed up to 4 weeks
  Measured in CORT-E2, FAST-3, IMV, IMV-ECLS domains
ICU and hospital free days | For FAST-3: ICU discharge, hospital discharge, Day 28. For IMPROV: Day 90.
  Measured in FAST-3, IMPROV domains
Discharge disposition. | Until hospital discharge, assessed up to 4 weeks
  Measured in IMV, IMV-ECLS, IMPROV domains. Location to which patient is discharged (e.g., home, weaning facility, etc.)
Days alive and at home to day 90 | Day 90
  Measured in IMV, IMV-ECLS and FLUDRO-1 domains
Need for ICU readmission prior to hospital discharge | Until hospital discharge, assessed up to 4 weeks
  Measured in IMV, IMV-ECLS domains
Duration of NIV | Until ICU discharge, typically within 28 days
  Measured in CORT-E2 domain
Duration of supplemental oxygen use | Until ICU discharge, typically within 28 days
  Measured in CORT-E2 domain
Need for ECLS | Until ICU discharge, typically within 28 days
  Measured in CORT-E2 domain
Duration of ECLS, only for patients who require ECLS | Until ICU discharge, typically within 28 days
  Measured in CORT-E2, IMV-ECLS domains.
Ventilator-free days until day 30 for CORT-E2, and until day 28 for FAST-3, FLUDRO-1 and ULTIMATE (an ordinal scale composed of survival to hospital discharge and days alive and free of ventilation where death in the hospital is assigned a score of -1). | Until day 30 for CORT-E2, and until day 28 for FAST-3, FLUDRO-1 and ULTIMATE
  Measured in CORT-E2, FAST-3, FLUDRO-1, and ULTIMATE domains.
EQ-5-D at day 180 | For CORT-E2, FAST-3, IMV, and IMV-ECLS domains: Day 180; For IMPROV domain: Day 90 and Day 180.
  Measured in CORT-E2, FAST-3, IMV, IMV-ECLS, IMPROV domains
Montreal Cognitive Assessment (MoCA) At day 180 | Day 180
  Measured in FAST-3 domain
Complications from corticosteroids. | Until hospital discharge, assessed up to 4 weeks
  Measured in CORT-E2 domain. Hypernatremia, hyperglycemia, delirium, clinically important GI bleeding, nosocomial infection, neuromuscular weakness.
  Measured in FLUDRO-1 domain: Hypernatremia, Hyperglycemia, Hypokalemia, Clinically important gastrointestinal bleeding, New nosocomial infection
Reintubation during index ICU admission | Until ICU discharge, typically within 28 days
  Measured in IMV, IMV-ECLS domains
Number of reintubations up to tracheostomy during index hospitalization | Until hospital discharge
  Measured in IMPROV domain
Tracheostomy during index ICU admission | Until ICU discharge, typically within 28 days
  Measured in IMV, IMV-ECLS, IMPROV domains
Re-cannulation to ECLS during index ICU admission | Until ICU discharge, typically within 28 days
  Measured in IMV-ECLS domain
Sequential Organ Failure Assessment (SOFA) score | Daily, for duration of intervention
  Measured in IMV, IMV-ECLS domains
Respiratory mechanics and gas exchange - Driving pressure. | Daily, for duration of intervention
  Measured in IMV, IMV-ECLS domains.
Respiratory mechanics and gas exchange - Pocc. | Daily, for duration of intervention
  Measured in IMV, IMV-ECLS domains.
Respiratory mechanics and gas exchange - P0.1 | Daily, for duration of intervention
  Measured in IMV, IMV-ECLS domains.
Respiratory mechanics and gas exchange - plateau airway pressure | Daily, for duration of intervention
  Measured in IMV, IMV-ECLS domains.
Respiratory mechanics and gas exchange - P/F ratio | Daily, for duration of intervention
  Measured in IMV, IMV-ECLS domains.
Respiratory mechanics and gas exchange - ventilatory ratio | Daily, for duration of intervention
  Measured in IMV domain.
Diaphragm thickness | Daily, for duration of intervention
  Measured in IMV domain
Maximal diaphragm thickening fraction | During first SBT
  Measured in IMV domain
Survival status at disconnection from mechanical ventilation (dead or alive) | Until day 28
  Measured in EXPAND-ECLS domain
Organ failure-free days | Until day 28
  Measured in ESCAPE, FLUDRO-1 domains
Serious adverse events (SAEs) | Throughout the trial
  Serious adverse events (SAEs) related to the intervention measured in FAST-3 domain
Modified Lung Injury Score (mLIS) | Until day 10
  Measured in IMV-EIT intervention. Calculated daily up until study day 10 in patients who are alive and continue to have acute hypoxemic respiratory failure requiring invasive mechanical ventilation.
Number of days from first SBT to disconnection from mechanical ventilation | Until ICU discharge
  Measured in IMPROV domain - final date of extubation or the first day of continuous tracheostomy mask for at least 24 hours, provided ventilator support is not resumed during the index ICU admission.
Barotrauma during hospital admission | Until 45 days or hospital discharge
  Measured in IMPROV domain including pneumothorax, pneumomediastinum, subcutaneous emphysema
Cardiac arrest during hospital admission | Until 45 days or hospital discharge
  Measured in IMPROV domain
30 second sit to stand test at ICU discharge and hospital discharge | Until ICU discharge, typically within 28 days
  Measured in IMPROV domain
Modified Medical Research Council (mMRC) Dyspnea Scale | At ICU discharge, Day 90, Day 180
  Measured in IMPROV domain
Physical function (Activity Measure for Post-Acute Care) | At ICU discharge, Day 90, Day 180
  Measured in IMPROV domain

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Goligher, MD, PhD, Study Chair — University Health Network, Toronto; Eddy Fan, MD, PhD, Study Chair — University Health Network, Toronto; Niall Ferguson, MD, MSc, Principal Investigator — University Health Network, Toronto; Lorenzo Del Sorbo, MD, Principal Investigator — University Health Network, Toronto; Bram Rochwerg, MD, MSc, Principal Investigator — McMaster University; Bijan Teja, MD, Principal Investigator — Unity Health Toronto; John Muscedere, MD, Principal Investigator — Queens University; Laveena Munshi, MD, Principal Investigator — Mount Sinai Hospital, Canada; Dmitry Rozenberg, MD, PhD, Principal Investigator — University Health Network, Toronto; Anastasia Newman, PhD, Principal Investigator — McMaster University
Locations (80):
- United States (24):
  - University of Arizona, Tucson, Arizona
  - University of California Los Angeles (UCLA), Los Angeles, California
  - University of San Diego (UCSD), San Diego, California
  - University of Colorado Hospital, Aurora, Colorado
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland Medical System, Baltimore, Maryland
  - The Johns Hopkins Medicine, Baltimore, Maryland
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - University of Michigan Health, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai New York City, New York, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Vanderbilt university medical center, Nashville, Tennessee
  - University of Utah Health, Farmington, Utah
  - Sentara Health, Norfolk, Virginia
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Flinders Medical Centre, Bedford Park, Southern Adelaide
  - St Vincents Sydney, Darlinghurst, Sydney
  - Bendigo Health Victoria, Bendigo, Victoria
  - University Hospital Geelong, Geelong, Victoria
  - The Austin Hospital, Heidelberg, Victoria
- Canada (35):
  - University of Calgary, Calgary, Alberta
  - University of Alberta/Edmonton University Hospital, Edmonton, Alberta
  - Nanaimo Regional General Hospital, Nanaimo, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Health Sciences Centre - Winnipeg, Winnipeg, Manitoba
  - Grace Hospital, Winnipeg, Manitoba
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - William Osler Health System, Brampton, Ontario
  - Brantford General Hospital, Brantford, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Oak Valley Health, Markham, Ontario
  - North York General Hospital, North York, Ontario
  - Lakeridge Hospital, Oshawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Ottawa Heart Research Institute, Ottawa, Ontario
  - Mackenzie Health, Richmond Hill, Ontario
  - Niagara Health Systems, Saint Catherines, Ontario
  - Scarborough Health Network, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Unity Health Toronto, Toronto, Ontario
  - Sinai Health, Mount Sinai Hospital, Toronto, Ontario
  - Cortellucci Vaughan Hospital, Vaughan, Ontario
  - Windsor Regional Health, Windsor, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - MUHC - McGill University Health Centre (Glen Site), Montreal, Quebec
  - Sacre Coeur du Montreal, Montreal, Quebec
  - Centre Hospitalier Universite de Sherbrooke, Sherbrooke, Quebec
  - Trois Riviere (CHAUR), Trois-Rivières, Quebec
  - Royal University Saskatoon, Saskatoon, Saskatchewan
  - University Health Network, Toronto
- Clínica Universidad de La Sabana, Chía, Cundinamarca, Colombia
- Italy (3):
  - Azienda Socio-Sanitaria Territoriale Ovest Milanese, Legnano, MI
  - Ospedale Maggiore, Fondazione IRCCS Ca Granda, Milano, Milan, MI
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
- New Zealand (4):
  - Auckland City Hospital, Grafton, Auckland
  - Middlemore Hospital, Auckland
  - Taranaki Base Hospital, New Plymouth
  - Rotorua Hospital, Rotorua
- King Abdulaziz Medical City- Riyadh, Riyadh, Saudi Arabia
- National University of Singapore, Singapore, Singapore
- Spain (3):
  - Parc Taulí University Hospital, Sabadell, Barcelona
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Josep Trueta (Girona), Girona